CLINICAL TRIAL: NCT06719817
Title: Evaluation of Some Trace Elements in Follicular Fluid in Intracytoplasmic Sperm Injection(ICSI) Patients
Brief Title: Evaluation of Some Trace Elements in Follicular Fluid in ICSI Cases and Their Effect on ICSI Outcomes
Acronym: ICSI
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Saad Waley, Doctor, Assiut University
Other Study IDs: AssiutU WHH
Record Dates: First submitted 2024-10-18; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Good Responders According to Guidelines Who Wre Charectarized by AMH>0.8ng/dl; Trace Elements in ICSI Cases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate concentrations of some trace elements in the follicular fluid and their reproductive outcomes.

DETAILED DESCRIPTION:
To evaluate some trace elements in the follicular fluid and their reproductive outcome

ELIGIBILITY:
Inclusion Criteria:good responders according to NICE guidelines with AMH more than 0.8ng/dl and antral follicular count more than 4 Exclusion Criteria:Poor responders according to ESHRE guidelines as advanced maternal age poor ovarian response and according to NICE guidelines AMH less than 0.8ng/dl

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: good responders according to NICE guidelines with AMH more than 0.8ng/dl and antral follicular count more than 4
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
oocyte maturity | 2024 to 2026
  Millimetres

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Egypt, Egypt